CLINICAL TRIAL: NCT02364323
Title: A Randomized Clinical Trial to Compare a Strategy Utilizing Genetic Testing and Personalized Risk Counseling With Standard Care on Patient Empowerment, Risk Factors Control and the Risk of Diabetic Complications
Brief Title: Genetic Testing and Counseling to Reduce Diabetic Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ronald C.W. Ma, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GEM Study
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Complication
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized risk counselling (Experimental): Intervention includes risk counseling to patients with diabetes on future risk of diabetic complications based on an established genetic counseling framework for common polygenic disorders which will be delivered to patient in a counselling sesssion 6 weeks after genetic testing
  Interventions: Behavioral: Personalized Risk Counselling
- Normal usual care (Placebo Comparator): Intervention includes normal usual care. General education on diabetes and diabetic complications
  Interventions: Other: Normal usual care

INTERVENTIONS:
Behavioral: Personalized Risk Counselling — Motivational message- towards lifestyle change, improved compliance and risk factors control Review overall control of clinical risk factors based on lab test results
  Arms: Personalized risk counselling
Other: Normal usual care — General education on diabetes and diabetic complications
  Arms: Normal usual care

SUMMARY:
The risk of diabetic kidney complications includes non-modifiable risk factors such as genetic predictors, as well as modifiable risk factors such as hyperglycaemia, hypertension, hyperlipidaemia and proteinuria. Genetic testing for personalized medicine is increasing in popularity, though evidence that genetic testing can empower patients to modify behaviour and reduce clinical risk remains lacking. In this project, the investigators aim to utilize a personalized risk counseling with genetic testing to evaluate its impact on risk factor control in diabetic patients. The investigators hypothesize that knowledge of genetic +/- clinical risk will empower patients and lead to improvement in the number of treatment targets achieved. The investigators will recruit 400 patients with diabetes. All subjects will undergo a comprehensive assessment of the risk of diabetic complications based on clinical risk factors. Half of the patients will be randomized to receive additional genetic testing of a panel of genetic markers proven to predict renal complications in our population: ACE I/D, aldose reductase (CA)n and PRKCB1 gene polymorphisms. The results of personalized risk assessment will be communicated by a health counsellor in the intervention arm. The impact of testing and patient knowledge of the result of genetic testing on achievement of treatment targets (A1c, BP, LDL-cholesterol, TG, use of ACEI/ARB) and patient behavior will be evaluated after 12 months. The other arm will receive results of the genetic testing at the completion of the study period. The study will help towards developing a strategy to empower patients through structured and personalized risk assessment will provide a novel approach to identify high-risk subjects for early intensive management, and may lead to reduction in long-term complications.

DETAILED DESCRIPTION:
Asia is in the midst of an epidemic of diabetes. Approximately 1 in 10 people in China has diabetes [1]. Asian patients with diabetes are characterized by early age of onset and increased risk of kidney complications. Young age of onset and long disease duration will place Chinese diabetic patients at high risk for complications. In the Hong Kong Diabetes Registry, which includes more than 7000 patients with type 2 diabetes, we have reported a high risk of diabetic complications, with 30% having died or sustained a major clinical event within 10years after diagnosis, including 10% developing cardiovascular complications, and 10% developing end-stage renal disease [2] [3]. The medical costs for the diabetic patient with complication is 2.2-3.8 fold that of patients without complications, and patients with cardiorenal complications are the most costly to manage [4]. Using our registry, we have identified clinical risk predictors for developing renal complications as glycaemic control, elevated blood pressure, hyperlipidaemia, and albuminuria [2] [3, 5], and have derived clinical risk prediction algorithms and incorporated them into a patient management portal, which can generate a standardized report for risk counseling based on clinical risk factors [6, 7]. Furthermore, in a multi-centre study utilizing a multidisciplinary team, we found that intensive management aiming to achieve targets of A1c, lipids, BP can significantly reduce the risk of developing kidney complication [8]. Therefore, the ability to identify subjects at risk of complications, and to target and motivate them to optimize modifiable risk factors for diabetic complications will be of clinical benefit and potentially cost-saving.

There has been much recent interest in the use of genetic testing for personalized medicine [9]. Diabetic kidney complications has high heritability of around 40% and several genetic factors have been found to be associated with diabetic renal complications. Using candidate-gene approach, our group has identified several genetic markers for diabetic kidney complications [10, 11] [12]. These include the angiotensin converting enzyme deletion/ insertion (ACE D/I) polymorphism and the aldose reductase (ALR2) 5'-(CA) n microsatellite polymorphism, each being associated with 2-3 fold increased risk of diabetic cardio-renal complications in Chinese [10, 13]. More recently, we have found that carriers of risk alleles at the protein kinase C-β1 (PRKCB1) locus can have up to 6-fold increased risk of developing end-stage renal disease during follow-up, after adjusting for the effect of clinical risk predictors [12].

The recent increase in consumer-initiated genetic testing has been driven by direct-to-consumer genetic testing, which assumes that personal genetic information can motivate positive behavioural change in patients [14]. Interestingly, a recent survey of patients without type 2 diabetes suggests that genetic testing may be able to motivate patients, with 71% of respondents reporting that they would be "much more motivated" to make behavioural changes if they were informed to be of high genetic risk for diabetes [15]. Although evidence that genetic testing can lead to behavioural changes is still lacking, several randomized clinical trials are currently underway to examine the impact of genetic testing on behaviour to reduce risk of diabetes. Given the disabling consequences of diabetic complications, and the ability to predict those at risk of developing complications, we plan to examine the role of personalized risk counseling incorporating genetic markers, and to examine its role in patient empowerment and risk factor control, which may help to reduce the risk of developing complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with type 2 diabetes aged 40-75 who can give informed consent
2. Subjects with no known chronic kidney disease (CKD defined as eGFR<60ml/min at baseline)
3. Suboptimal glucose control with HbA1c ≥ 7.5%
4. Known history of hypertension including elevated BP ≥140/90 on more than one occasion

Exclusion Criteria:

1. Subjects with known coronary artery disease or coronary revascularisation
2. Subjects with previous history of cerebrovascular accident
3. Subjects with known proliferative retinopathy or previous laser treatment for diabetic retinopathy
4. Subjects with life-threatening conditions including malignancy
5. Subjects with known psychiatric conditions including depression
6. Subjects with significant renal impairment (eGFR<60ml/min at baseline) or non-diabetic renal disease (e.g. biopsy-proven glomerulonephritis or obstructive uropathy)
7. Subjects with major physical disability

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
percentage of patients attaining ≥ 3 pre-defined treatment targets from the following treatment targets: 1) BP <130/80 mm Hg 2) HbA1c <7% 3) Calculated LDL-cholesterol <2.6mmol/l 4) Fasting TG <2mmol/l 5) Use of ACEI or ARB | At 1 year
  primary outcome of 3 out of 5 targets achieved as defined above

SECONDARY OUTCOMES:
microalbuminuria as a marker of degree of renal damage | At 1 year
  new onset of microalbuminuria at 1 year follow-up
Patient empowerment as measured on the Chinese Diabetes Empowerment Scale (DES) | At 1 year
  Score on the DES
Patient behavior measured on the Summary of Diabetes Self-care Activities (SDSCA) | At 1 year
  Score of diabetes self-care as measured by the SDSCA

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C Ma, MB BChir, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Yang W, Lu J, Weng J, Jia W, Ji L, Xiao J, Shan Z, Liu J, Tian H, Ji Q, Zhu D, Ge J, Lin L, Chen L, Guo X, Zhao Z, Li Q, Zhou Z, Shan G, He J; China National Diabetes and Metabolic Disorders Study Group. Prevalence of diabetes among men and women in China. N Engl J Med. 2010 Mar 25;362(12):1090-101. doi: 10.1056/NEJMoa0908292. PMID 20335585
- [Background] Chan JC, So W, Ma RC, Tong PC, Wong R, Yang X. The Complexity of Vascular and Non-Vascular Complications of Diabetes: The Hong Kong Diabetes Registry. Curr Cardiovasc Risk Rep. 2011 Jun;5(3):230-239. doi: 10.1007/s12170-011-0172-6. Epub 2011 Apr 12. PMID 21654912
- [Background] Yang XL, So WY, Kong AP, Clarke P, Ho CS, Lam CW, Ng MH, Lyu RR, Yin DD, Chow CC, Cockram CS, Tong PC, Chan JC. End-stage renal disease risk equations for Hong Kong Chinese patients with type 2 diabetes: Hong Kong Diabetes Registry. Diabetologia. 2006 Oct;49(10):2299-308. doi: 10.1007/s00125-006-0376-3. Epub 2006 Aug 30. PMID 16944095
- [Background] Chan BS, Tsang MW, Lee VW, Lee KK. Cost of Type 2 Diabetes mellitus in Hong Kong Chinese. Int J Clin Pharmacol Ther. 2007 Aug;45(8):455-68. doi: 10.5414/cpp45455. PMID 17725179
- [Background] Luk AO, So WY, Ma RC, Kong AP, Ozaki R, Ng VS, Yu LW, Lau WW, Yang X, Chow FC, Chan JC, Tong PC; Hong Kong Diabetes Registry. Metabolic syndrome predicts new onset of chronic kidney disease in 5,829 patients with type 2 diabetes: a 5-year prospective analysis of the Hong Kong Diabetes Registry. Diabetes Care. 2008 Dec;31(12):2357-61. doi: 10.2337/dc08-0971. Epub 2008 Oct 3. PMID 18835954
- [Background] Chan J, So W, Ko G, Tong P, Yang X, Ma R, Kong A, Wong R, Le Coguiec F, Tamesis B, Wolthers T, Lyubomirsky G, Chow P. The Joint Asia Diabetes Evaluation (JADE) Program: a web-based program to translate evidence to clinical practice in Type 2 diabetes. Diabet Med. 2009 Jul;26(7):693-9. doi: 10.1111/j.1464-5491.2009.02751.x. PMID 19573118
- [Background] Ko GT, So WY, Tong PC, Le Coguiec F, Kerr D, Lyubomirsky G, Tamesis B, Wolthers T, Nan J, Chan J. From design to implementation--the Joint Asia Diabetes Evaluation (JADE) program: a descriptive report of an electronic web-based diabetes management program. BMC Med Inform Decis Mak. 2010 May 13;10:26. doi: 10.1186/1472-6947-10-26. PMID 20465815
- [Background] Chan JC, So WY, Yeung CY, Ko GT, Lau IT, Tsang MW, Lau KP, Siu SC, Li JK, Yeung VT, Leung WY, Tong PC; SURE Study Group. Effects of structured versus usual care on renal endpoint in type 2 diabetes: the SURE study: a randomized multicenter translational study. Diabetes Care. 2009 Jun;32(6):977-82. doi: 10.2337/dc08-1908. PMID 19460913
- [Background] Malandrino N, Smith RJ. Personalized medicine in diabetes. Clin Chem. 2011 Feb;57(2):231-40. doi: 10.1373/clinchem.2010.156901. Epub 2010 Dec 2. PMID 21127150
- [Background] Wang Y, Ng MC, So WY, Tong PC, Ma RC, Chow CC, Cockram CS, Chan JC. Prognostic effect of insertion/deletion polymorphism of the ace gene on renal and cardiovascular clinical outcomes in Chinese patients with type 2 diabetes. Diabetes Care. 2005 Feb;28(2):348-54. doi: 10.2337/diacare.28.2.348. PMID 15677791
- [Background] Wang Y, Luk AO, Ma RC, So WY, Tam CH, Ng MC, Yang X, Lam V, Tong PC, Chan JC. Predictive role of multilocus genetic polymorphisms in cardiovascular disease and inflammation-related genes on chronic kidney disease in Type 2 diabetes--an 8-year prospective cohort analysis of 1163 patients. Nephrol Dial Transplant. 2012 Jan;27(1):190-6. doi: 10.1093/ndt/gfr343. Epub 2011 Jul 15. PMID 21765051
- [Background] Ma RC, Tam CH, Wang Y, Luk AO, Hu C, Yang X, Lam V, Chan AW, Ho JS, Chow CC, Tong PC, Jia W, Ng MC, So WY, Chan JC. Genetic variants of the protein kinase C-beta 1 gene and development of end-stage renal disease in patients with type 2 diabetes. JAMA. 2010 Aug 25;304(8):881-9. doi: 10.1001/jama.2010.1191. PMID 20736472
- [Background] So WY, Wang Y, Ng MC, Yang X, Ma RC, Lam V, Kong AP, Tong PC, Chan JC. Aldose reductase genotypes and cardiorenal complications: an 8-year prospective analysis of 1,074 type 2 diabetic patients. Diabetes Care. 2008 Nov;31(11):2148-53. doi: 10.2337/dc08-0712. Epub 2008 Aug 20. PMID 18716049
- [Background] Janssens AC, Gwinn M, Bradley LA, Oostra BA, van Duijn CM, Khoury MJ. A critical appraisal of the scientific basis of commercial genomic profiles used to assess health risks and personalize health interventions. Am J Hum Genet. 2008 Mar;82(3):593-9. doi: 10.1016/j.ajhg.2007.12.020. PMID 18319070
- [Background] Grant RW, Hivert M, Pandiscio JC, Florez JC, Nathan DM, Meigs JB. The clinical application of genetic testing in type 2 diabetes: a patient and physician survey. Diabetologia. 2009 Nov;52(11):2299-2305. doi: 10.1007/s00125-009-1512-7. Epub 2009 Sep 2. PMID 19727660
- [Background] Chen S, Chiu H, Xu B, Ma Y, Jin T, Wu M, Conwell Y. Reliability and validity of the PHQ-9 for screening late-life depression in Chinese primary care. Int J Geriatr Psychiatry. 2010 Nov;25(11):1127-33. doi: 10.1002/gps.2442. PMID 20029795
- [Background] Ting RZ, Nan H, Yu MW, Kong AP, Ma RC, Wong RY, Loo K, So WY, Chow CC, Ko GT, Wing YK, Chan JC. Diabetes-related distress and physical and psychological health in chinese type 2 diabetic patients. Diabetes Care. 2011 May;34(5):1094-6. doi: 10.2337/dc10-1612. Epub 2011 Mar 11. PMID 21398526
- [Background] Shiu AT, Martin CR, Thompson DR, Wong RY. Psychometric properties of the Chinese version of the diabetes empowerment scale. Psychol Health Med. 2006 May;11(2):198-208. doi: 10.1080/13548500500286845. PMID 17129908